CLINICAL TRIAL: NCT07058532
Title: Therapeutic Writing Intervention in Pain Rehabilitation
Brief Title: Therapeutic Writing for Adults Suffering From Chronic Pain and Comorbid Mental Health Disorders
Acronym: TWfCP&MH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toni Salikka (Other)
Responsible Party: Sponsor-Investigator, Toni Salikka, MA, PhD Candidate, Tampere University
Organization: Tampere University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R25034
Record Dates: First submitted 2025-06-23; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain; Mental Health Disorder; Psychiatric &Amp;Amp;or Mood Disorder; Psychiatric Comorbidities; Psychiatric Diagnosis; Emotional Pain; Emotional Distress; Emotion Regulation; Emotional Processing; Meaning of Life; Meaning Made; Meaning of Life and Life Satisfaction; Depressive Disorder; Anxiety Disorders; Sleep Disorder; Comorbid Depression; Process, Acceptance
Keywords: Therapeutic writing; Chronic pain; Mental health disorders; Psychiatric disorders; Emotion regulation; Emotional processing; Meaning-making; Non-pharmacological intervention; Logotherapy; Phenomenological analysis; Psychosocial rehabilitation; Pain management; Pain coping; Creative writing
MeSH Terms: conditions — Chronic Pain; Mental Disorders; Emotional Regulation; Personal Satisfaction; Depressive Disorder; Anxiety Disorders; Sleep Wake Disorders; Behavior; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic Writing Intervention in Pain Rehabilitation (Experimental): Participants in this single-arm study will take part in a structured therapeutic writing intervention as part of a multidisciplinary pain rehabilitation program at the Pain Clinic of Satasairaala Hospital. The study spans approximately three months and includes around 11 clinic visits. The intervention is delivered in two phases: first, four consecutive daily writing sessions (20 minutes each), followed by four weekly sessions (30-60 minutes each). Prior to the intervention, participants are assessed for eligibility by the clinic's multidisciplinary team and interviewed by the principal investigator. Post-intervention, participants are interviewed twice to explore their health-related experiences with the writing process.
  Interventions: Other: Therapeutic Writing Intervention in Pain Rehabilitation

INTERVENTIONS:
Other: Therapeutic Writing Intervention in Pain Rehabilitation — The therapeutic writing intervention is designed to support emotional processing and regulation in individuals with chronic pain and comorbid mental health disorders. It has been developed specifically for use in a clinical rehabilitation setting and is delivered in two phases over a four-week period at the Pain Clinic of Satasairaala Hospital. Sessions are conducted in person, with clinical staff available to support participants. The intervention is non-pharmacological, low-risk, and integrated into the broader multidisciplinary care pathway.

SUMMARY:
The goal of this observational study is to understand the effects and experiences of therapeutic writing interventions in adult women with chronic pain and co-occurring mental health conditions. The main questions it aims to answer are:

Can therapeutic writing help relieve chronic pain and emotional distress?

How does writing support emotional processing, regulation, and meaning-making during rehabilitation?

Participants will take part in a two-part writing intervention involving:

Guided writing exercises that focus on emotional processing, emotion regulation, and creating meaning.

Individual interviews after the writing sessions to explore their experiences.

The study uses qualitative analysis methods-phenomenology and logotherapy-to better understand how these writing interventions may support recovery, improve well-being, and offer non-pharmacological tools for managing chronic pain and mental health challenges.

DETAILED DESCRIPTION:
Chronic pain affects approximately 20% of the global population and represents one of the most widespread causes of disability worldwide. Individuals living with chronic pain often experience additional mental health challenges-such as depression, anxiety, or trauma-related disorders-which compound their suffering and reduce quality of life. Traditional pain management strategies often focus on physical symptoms, while the emotional and psychological dimensions may remain under-addressed.

This study aims to explore the potential of therapeutic writing-a psychological intervention that encourages participants to express and process emotions through guided writing exercises-as a complementary approach for improving health and well-being in individuals with both chronic pain and mental health conditions.

The study is being conducted at the Department of Physical Medicine and Rehabilitation of Satasairaala Hospital in Finland and involves five adult female participants with chronic pain and comorbid psychiatric conditions. Each participant will engage in a two-part writing intervention that incorporates techniques grounded in emotional processing, emotion regulation, and meaning-making. These exercises are designed to help individuals articulate their internal experiences, explore the personal impact of pain and illness, and foster a sense of psychological coherence.

Data collection spans two sub-studies:

Sub-studies 1 and 2 involve qualitative interviews with participants following the intervention, capturing their firsthand experiences and perceived effects.

The qualitative data will be analyzed using a multi-method approach, combining phenomenological analysis-which highlights the participants' lived experiences-and logotherapy-informed analysis, which examines how therapeutic writing supports the search for meaning during rehabilitation. This dual approach provides a comprehensive view of how narrative expression may influence recovery pathways.

The ultimate goal is to identify writing-based strategies that can complement clinical care for this patient population and inform future updates to rehabilitation programs and treatment guidelines-both locally and nationally. If proven beneficial, therapeutic writing could serve as an accessible, cost-effective, and non-pharmacological tool to enhance holistic pain care and mental health support.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (18 years or older), assigned female at birth and self-identify as women
* Diagnosed with or experience of chronic, widespread (non-cancer) pain lasting at least two years
* Diagnosed with or living with one or more mild mental health disorders (e.g., anxiety, mild depression), without current or past severe psychiatric conditions
* Diagnosed with or experience of nociplastic pain (e.g., fibromyalgia)
* Not currently using medications that may impair cognitive functioning (e.g., benzodiazepines, anticholinergics, opioids, antipsychotics)
* Able to attend approximately 11 in-person visits over a 3-month period
* Willing and able to participate in a structured therapeutic writing intervention
* Purposefully selected to reflect a range of lived experiences relevant to the study's aims

Exclusion Criteria:

* Presence of severe mental health disorders (e.g., schizophrenia, bipolar disorder, severe depression, or other psychotic conditions)
* Use of medications known to impair memory, attention, or decision-making (e.g., benzodiazepines, anticholinergics, opioids, antipsychotics)
* Participation in other concurrent treatments that may influence study outcomes
* Cognitive limitations that would hinder meaningful engagement in the writing intervention
* Individuals not assigned female at birth or who do not identify as women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals who self-identify as women and were assigned female at birth are eligible to participate.
Enrollment: 5 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Health-Related Experiences of Participants | Baseline (prior to intervention), immediately post-intervention (Week 5), and 3 months post-intervention (Week 17)
  Description:
  Qualitative themes identified from semi-structured interviews exploring participants' perceived health-related changes following the writing intervention, including emotional processing, emotion regulation, and meaning-making.
  Unit of Measure:
  Thematic categories derived from qualitative content analysis.
  Time Frame:
  Data will be collected through semi-structured interviews conducted at three time points: prior to the writing intervention (baseline), immediately after the final writing session (Week 5), and three months after the intervention (Week 17).

SECONDARY OUTCOMES:
Perceived Impact on Emotion Regulation | Baseline (prior to intervention), immediately post-intervention (Week 5), and 3 months post-intervention (Week 17)
  Participant-reported changes in emotional awareness, expression, and regulation, identified through qualitative analysis of semi-structured interviews conducted immediately post-intervention.
  Original Unit of Measure: Thematic categories and frequency of emotion regulation-related content identified through qualitative content analysis.
  Time Frame: Data will be collected through semi-structured interviews conducted at three time points: prior to the writing intervention (baseline), immediately after the final writing session (Week 5), and three months after the intervention (Week 17).
Themes of Meaning-Making and Future Orientation Identified Through Qualitative Interview Analysis | Baseline (prior to intervention), immediately post-intervention (Week 5), and 3 months post-intervention (Week 17)
  Description:
  Themes related to personal meaning, future goals, and psychological growth will be assessed through qualitative content analysis of semi-structured interviews conducted at three time points: baseline, immediately post-intervention (Week 5), and 3 months post-intervention (Week 17).
  Unit of Measure:
  Thematic categories and depth of meaning-making and future orientation content identified through qualitative content analysis.
  Time Frame:
  Baseline (prior to intervention), immediately post-intervention (Week 5), and 3 months post-intervention (Week 17)

CONTACTS AND LOCATIONS:
Locations (1):
- Satasairaala Hospital, Department of Physical Medicine and Rehabilitation: Pain Clinic, Pori, Satakunta, Finland

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy and confidentiality concerns. The data includes sensitive personal information that cannot be fully anonymized without risking participant identification.